CLINICAL TRIAL: NCT02365636
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Topically Applied TV-45070 (4% and 8% w/w Ointment) in Patients With Postherpetic Neuralgia.
Brief Title: A Study to Evaluate the Safety and Efficacy of Topically Applied TV 45070 Ointment in Patients With Postherpetic Neuralgia (PHN)
Acronym: (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TV-45070-CNS-20013
Record Dates: First submitted 2015-02-13; First posted 2015-02-19 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — TV-45070

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TV-45070 4% (Experimental): TV-45070 ointment in a 4% strength applied topically twice daily to the area of postherpetic neuralgia (PHN) pain during the treatment period from days 1 through 28.
  Interventions: Drug: TV-45070
- TV-45070 8% (Experimental): TV-45070 ointment in a 8% strength applied topically twice daily to the area of postherpetic neuralgia (PHN) pain during the treatment period from days 1 through 28.
  Interventions: Drug: TV-45070
- Placebo (Placebo Comparator): Placebo ointment applied topically twice daily to the area of postherpetic neuralgia (PHN) pain during the treatment period from days 1 through 28.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TV-45070 — TV-45070 is an ointment applied topically twice daily to area of pain.
  Other Names: funapide; XEN402
  Arms: TV-45070 4%; TV-45070 8%
Drug: Placebo — The matching placebo ointment contained only the excipients of the active treatment; also applied topically twice daily to area of pain.
  Arms: Placebo

SUMMARY:
This is a study to evaluate the safety and efficacy of 4% and 8% w/w TV 45070 ointment compared with placebo ointment applied topically and twice daily to the area of PHN pain for 4 weeks in patients with PHN

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic Postherpetic Neuralgia (PHN), defined as pain present for more than 6 months and less than 10 years after onset of herpes zoster skin rash affecting a single dermatome. Patients with more than 1 involved dermatome may also be included, provided the affected dermatomes are contiguous.
* Patient is ≥18 years of age, with a body mass index (BMI) between 18 and 34 kg/m2, inclusive, at the screening visit.
* If the patient is a woman and is fertile, the patient is not pregnant and has negative pregnancy tests at both the screening and randomization visits, and agrees to use an acceptable method of contraception for the duration of the study, including follow-up.
* If the patient is a man and is capable of producing offspring, the patient must agree to use an acceptable method of contraception, unless the partner cannot become pregnant for the duration of the study, including follow-up.
* Patient must sign the written Informed Consent Form (ICF) for the study and be willing to comply with all study procedures and restrictions.
* Patient must be judged by the investigator to be medically healthy (except for PHN) and able to participate in the study

  * Other criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Patient has any other severe pain that might confound assessment or self-evaluation of pain due to PHN.
* Patient has PHN affecting the face (trigeminal nerve distribution).
* Patient has a history, in the judgment of the investigator, of inadequate response to more than 3 adequate courses of treatment with other medications used to treat neuropathic pain (eg, tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitors, anticonvulsants, topical lidocaine, and/or topical capsaicin).
* Patient is taking oral analgesics (either opioid or non-opioid) or is receiving topical therapy such as the 5% topical lidocaine patch for the treatment of pain and is unwilling or unable to complete a washout period during which the patient will discontinue analgesic therapy or topical pain therapy.
* Patient has been treated with topical capsaicin at any time in the past 6 months for neuropathic pain.
* Patient has a history of fibromyalgia.

  * Other criteria apply, please contact the investigator for more information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (77):
- United States (77):
  - Teva Investigational Site 13052, Birmingham, Alabama
  - Teva Investigational Site 13086, Mobile, Alabama
  - Teva Investigational Site 13514, Phoenix, Arizona
  - Teva Investigational Site 13520, Phoenix, Arizona
  - Teva Investigational Site 13661, Little Rock, Arkansas
  - Teva Investigational Site 13079, Colton, California
  - Teva Investigational Site 13331, Pomona, California
  - Teva Investigational Site 13341, Sacramento, California
  - Teva Investigational Site 13051, Santa Monica, California
  - Teva Investigational Site 13055, Thousand Oaks, California
  - Teva Investigational Site 13100, Torrance, California
  - Teva Investigational Site 13657, Milford, Connecticut
  - Teva Investigational Site 13521, Brandon, Florida
  - Teva Investigational Site 13085, Brooksville, Florida
  - Teva Investigational Site 13057, Clearwater, Florida
  - Teva Investigational Site 13084, Fort Myers, Florida
  - Teva Investigational Site 13047, Hialeah, Florida
  - Teva Investigational Site 13046, Homestead, Florida
  - Teva Investigational Site 13098, Jacksonville, Florida
  - Teva Investigational Site 13045, Kissimmee, Florida
  - Teva Investigational Site 13064, Miami, Florida
  - Teva Investigational Site 13338, Miami, Florida
  - Teva Investigational Site 13044, Miami, Florida
  - Teva Investigational Site 13335, Miami, Florida
  - Teva Investigational Site 13522, Naples, Florida
  - Teva Investigational Site 13058, New Port Richey, Florida
  - Teva Investigational Site 13076, Oldsmar, Florida
  - Teva Investigational Site 13073, Orlando, Florida
  - Teva Investigational Site 13048, Orlando, Florida
  - Teva Investigational Site 13659, Pembroke Pines, Florida
  - Teva Investigational Site 13519, Seminole, Florida
  - Teva Investigational Site 13056, St. Petersburg, Florida
  - Teva Investigational Site 13059, Tampa, Florida
  - Teva Investigational Site 13329, Venice, Florida
  - Teva Investigational Site 13513, Virginia Gardens, Florida
  - Teva Investigational Site 13053, Atlanta, Georgia
  - Teva Investigational Site 13063, Marietta, Georgia
  - Teva Investigational Site 13091, Aurora, Illinois
  - Teva Investigational Site 13072, Bolingbrook, Illinois
  - Teva Investigational Site 13062, Evansville, Indiana
  - Teva Investigational Site 13093, Evansville, Indiana
  - Teva Investigational Site 13074, Monroe, Louisiana
  - Teva Investigational Site 13660, Shreveport, Louisiana
  - Teva Investigational Site 13094, Brockton, Massachusetts
  - Teva Investigational Site 13061, Detroit, Michigan
  - Teva Investigational Site 13049, Farmington Hills, Michigan
  - Teva Investigational Site 13099, St Louis, Missouri
  - Teva Investigational Site 13065, Las Vegas, Nevada
  - Teva Investigational Site 13066, Albuquerque, New Mexico
  - Teva Investigational Site 13330, Albuquerque, New Mexico
  - Teva Investigational Site 13658, Albany, New York
  - Teva Investigational Site 13334, Brooklyn, New York
  - Teva Investigational Site 13054, New York, New York
  - Teva Investigational Site 13083, North Massapequa, New York
  - Teva Investigational Site 13060, Calabash, North Carolina
  - Teva Investigational Site 13337, Raleigh, North Carolina
  - Teva Investigational Site 13082, Winston-Salem, North Carolina
  - Teva Investigational Site 13089, Columbus, Ohio
  - Teva Investigational Site 13075, Oklahoma City, Oklahoma
  - Teva Investigational Site 13328, Oklahoma City, Oklahoma
  - Teva Investigational Site 13516, Oklahoma City, Oklahoma
  - Teva Investigational Site 13078, Eugene, Oregon
  - Teva Investigational Site 13333, Levittown, Pennsylvania
  - Teva Investigational Site 13339, Philadelphia, Pennsylvania
  - Teva Investigational Site 13327, Pittsburgh, Pennsylvania
  - Teva Investigational Site 13332, Charleston, South Carolina
  - Teva Investigational Site 13068, Rapid City, South Dakota
  - Teva Investigational Site 13095, Knoxville, Tennessee
  - Teva Investigational Site 13096, Memphis, Tennessee
  - Teva Investigational Site 13070, Arlington, Texas
  - Teva Investigational Site 13088, Austin, Texas
  - Teva Investigational Site 13340, McKinney, Texas
  - Teva Investigational Site 13050, Plano, Texas
  - Teva Investigational Site 13518, Salt Lake City, Utah
  - Teva Investigational Site 13090, Norfolk, Virginia
  - Teva Investigational Site 13081, Bellevue, Washington
  - Teva Investigational Site 13336, Seattle, Washington

REFERENCES:
- [Derived] Fetell M, Sendel M, Li T, Marinelli L, Vollert J, Ruggerio E, Houk G, Dockum M, Albrecht PJ, Rice FL, Baron R. Cutaneous nerve fiber and peripheral Nav1.7 assessment in a large cohort of patients with postherpetic neuralgia. Pain. 2023 Nov 1;164(11):2435-2446. doi: 10.1097/j.pain.0000000000002950. Epub 2023 Jun 27. PMID 37366590

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 658 patients with chronic postherpetic neuralgia (PHN) were screened; reasons for not enrolling included: inclusion criteria not met (144), exclusion criteria met (171), consent withdrawn (28), lost to follow-up (6), adverse event (1), other (8).
Pre-assignment Details: 300 participants were randomly assigned in a 1:1:1 ratio to 1 of 3 treatment groups.
Period: Overall Study
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Started | 100 | 100 | 100
Safety Population | 100 | 98 (2 terminated prior to treatment due to 1) prohibited concomitant medication 2) exclusion criteria) | 100
Full Analysis Set | 100 | 98 | 100
Completed | 94 | 93 | 97
Not Completed | 6 | 7 | 3
Not completed — Adverse Event | 3 | 3 | 2
Not completed — Protocol Violation | 1 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (15.99) | 57.6 (16.61) | 58.6 (15.80) | 57.8 (16.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 50 | 65 | 172
  Male | 43 | 50 | 35 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 53 | 70 | 179
  Not Hispanic or Latino | 43 | 47 | 30 | 120
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 81 | 79 | 90 | 250
  Black or African American | 13 | 17 | 7 | 37
  Asian | 3 | 3 | 1 | 7
  American Indian or Alaskan Native | 1 | 1 | 1 | 3
  Other | 2 | 0 | 1 | 3
Weight [Mean (Standard Deviation); unit: kg] | 77.02 (13.775) | 77.41 (13.383) | 77.86 (15.111) | 77.43 (14.066)
Height [Mean (Standard Deviation); unit: cm] | 167.27 (10.258) | 168.03 (8.203) | 165.82 (10.355) | 167.04 (9.668)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.42 (3.457) | 27.30 (3.452) | 28.15 (3.798) | 27.62 (3.580)
R1150W Polymorphism Status [Count of Participants; unit: Participants] — Patients who carry the R1150W polymorphism have a nucleotide containing adenine (A) instead of guanine (G) in the rs6746030 single nucleotide polymorphism in the SCN9A gene. This change causes an arginine to tryptophan amino acid residue change at position 1150 in the alpha subunit of the voltage-gated sodium channel NaV1.7. Those who carry the R1150W polymorphism may be heterozygous (GA) or homozygous (AA) for the minor allele. This R1150W polymorphism in the SCN9A gene may affect pain perception (Reimann et al 2010).
  Participants
    Homozygous minor allele (positive, AA) | 1 | 2 | 0 | 3
    Heterozygous (positive, AG) | 17 | 25 | 22 | 64
    Homozygous common allele (negative, GG) | 82 | 73 | 78 | 233

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in the Weekly Average of the Daily Average Numeric Rating Scale (NRS) Pain Scores Using a Mixed Model for Repeated Measures
Description: The primary efficacy endpoint was the change from baseline to week 4 in the weekly average of the daily average NRS scores. The NRS is a widely-used, standard one-dimensional 11-point scale from 0=no pain to 10=worst pain imaginable as reported by patients. The daily average NRS scores is the average of the 2 NRS scores (recorded in the morning and evening) of average pain, defined as the patient-reported average pain intensity over the prior 12 hours. At least 1 of the 2 daily scores had to be recorded (non-missing) or the daily average was considered missing. Negative change from baseline values indicate a lessening of pain. The Mixed Model Repeated Measures (MMRM) model with change from baseline in the weekly average of the daily average NRS scores at week 4 as the dependent variable; week, pooled study center, treatment, and treatment by visit interaction as fixed factors, baseline weekly average of the daily average NRS scores as covariate; and patient as a random effect.
Time Frame: Baseline (day -7 to day -1), Week 4 (day 22 to day 28)
Population: Full analysis set; patients from one site are excluded due to lack of data integrity.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
units on a scale
  Baseline: number analyzed (Participants) | 98 | 98 | 100
  Baseline | 5.37 (0.992) | 5.60 (1.236) | 5.51 (0.963)
  Change from baseline at week 4: number analyzed (Participants) | 94 | 93 | 97
  Change from baseline at week 4 | -1.64 (1.360) | -1.71 (1.500) | -1.90 (1.670)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; The Mixed Model Repeated Measures (MMRM) model with change from baseline in the weekly average of the daily average NRS scores at week 4 as the dependent variable; week, pooled study center, treatment, and treatment by visit interaction as fixed factors, baseline weekly average of the daily average NRS scores as covariate; and patient as a random effect; Test type: Superiority; p = 0.130, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.32, 95% CI 2-sided [-0.094 to 0.726]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.245, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.24, 95% CI 2-sided [-0.167 to 0.652]

2. Secondary Outcome: Change From Baseline to Week 4 in the Weekly Average of the Average Numeric Rating Scale (NRS) Pain Scores Recorded in the Evening Using a Mixed Model for Repeated Measures
Description: The NRS is a widely-used, standard one-dimensional 11-point scale from 0=no pain to 10=worst pain imaginable as reported by patients. The NRS pain scores recorded in the evening is defined as the patient-reported average pain intensity over the prior 12 hours. Negative change from baseline values indicate a lessening of pain. The Mixed Model Repeated Measures (MMRM) model with change from baseline in the weekly average of the evening NRS scores at week 4 as the dependent variable; week, pooled study center, treatment, and treatment by visit interaction as fixed factors, baseline weekly average of the evening NRS scores as covariate; and patient as a random effect.
Time Frame: Baseline (day -7 to day -1), Week 4 (day 22 to day 28)
Population: Full analysis set. Participants from one site are excluded due to lack of data integrity.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
units on a scale
  Baseline: number analyzed (Participants) | 98 | 98 | 100
  Baseline | 5.45 (1.073) | 5.66 (1.320) | 5.58 (0.994)
  Change from baseline at week 4: number analyzed (Participants) | 94 | 93 | 97
  Change from baseline at week 4 | -1.70 (1.412) | -1.73 (1.506) | -1.96 (1.745)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; The Mixed Model Repeated Measures (MMRM) model with change from baseline in the weekly average of the average NRS pain scores recorded in the evening at week 4 as the dependent variable; week, pooled study center, treatment, and treatment by visit interaction as fixed factors, baseline weekly average of the average NRS pain scores recorded in the evening as covariate; and patient as a random effect; Test type: Superiority; p = 0.128, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.32, 95% CI 2-sided [-0.093 to 0.735]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.194, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.27, 95% CI 2-sided [-0.140 to 0.688]

3. Secondary Outcome: Change From Baseline to Week 4 in the Weekly Average of the Average Numeric Rating Scale (NRS) Pain Scores Recorded in the Morning Using a Mixed Model for Repeated Measures
Description: The NRS is a widely-used, standard one-dimensional 11-point scale from 0=no pain to 10=worst pain imaginable as reported by patients. The NRS pain scores recorded in the morning is defined as the patient-reported average pain intensity over the prior 12 hours. Negative change from baseline values indicate a lessening of pain. The Mixed Model Repeated Measures (MMRM) model with change from baseline in the weekly average of the evening NRS scores at week 4 as the dependent variable; week, pooled study center, treatment, and treatment by visit interaction as fixed factors, baseline weekly average of morning NRS scores as covariate; and patient as a random effect.
Time Frame: Baseline (day -7 to day -1), Week 4 (day 22 to day 28)
Population: Full analysis set. Participants from one site are excluded due to lack of data integrity.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
units on a scale
  Baseline: number analyzed (Participants) | 98 | 98 | 100
  Baseline | 5.30 (0.980) | 5.53 (1.226) | 5.44 (0.968)
  Change from baseline at week 4: number analyzed (Participants) | 94 | 93 | 97
  Change from baseline at week 4 | -1.60 (1.386) | -1.68 (1.548) | -1.84 (1.623)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; The Mixed Model Repeated Measures (MMRM) model with change from baseline in the weekly average of the average NRS pain scores recorded in the morning at week 4 as the dependent variable; week, pooled study center, treatment, and treatment by visit interaction as fixed factors, baseline weekly average of the average NRS pain scores recorded in the morning as covariate; and patient as a random effect; Test type: Superiority; p = 0.177, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.28, 95% CI 2-sided [-0.128 to 0.691]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.325, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.20, 95% CI 2-sided [-0.204 to 0.614]

4. Secondary Outcome: Change From Baseline to Week 4 in the Weekly Average of the Worst Numeric Rating Scale (NRS) Pain Scores Recorded in the Evening Using a Mixed Model for Repeated Measures
Description: The NRS is a widely-used, standard one-dimensional 11-point scale from 0=no pain to 10=worst pain imaginable as reported by patients. The worst pain is defined as the patient-reported worst pain intensity over the prior 24 hours. Negative change from baseline values indicate a lessening of pain. The Mixed Model Repeated Measures (MMRM) model with change from baseline in the weekly average of the worst pain NRS scores at week 4 as the dependent variable; week, pooled study center, treatment, and treatment by visit interaction as fixed factors, baseline weekly average of the evening NRS scores as covariate; and patient as a random effect.
Time Frame: Baseline (day -7 to day -1), Week 4 (day 22 to day 28)
Population: Full analysis set. Participants from one site are excluded due to lack of data integrity.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
units on a scale
  Baseline: number analyzed (Participants) | 98 | 98 | 100
  Baseline | 6.09 (1.060) | 6.35 (1.378) | 6.09 (1.041)
  Change from baseline at week 4: number analyzed (Participants) | 94 | 93 | 97
  Change from baseline at week 4 | -1.73 (1.576) | -1.83 (1.657) | -1.97 (1.883)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; The Mixed Model Repeated Measures (MMRM) model with change from baseline in the weekly average of the worst NRS pain scores recorded in the evening at week 4 as the dependent variable; week, pooled study center, treatment, and treatment by visit interaction as fixed factors, baseline weekly average of the worst NRS pain scores recorded in the evening as covariate; and patient as a random effect; Test type: Superiority; p = 0.202, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.29, 95% CI 2-sided [-0.158 to 0.741]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.457, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.457, 95% CI 2-sided [-0.280 to 0.621]

5. Secondary Outcome: Percentage of Participants With >=30% and >=50% Improvement From Baseline in the Weekly Average of the Daily Average Numeric Rating Scale (NRS) Pain Scores at Week 4 Using a Mixed Model for Repeated Measures
Description: The NRS is a 11-point scale from 0=no pain to 10=worst pain imaginable as reported by patients. The daily average NRS scores is the average of the 2 NRS scores (recorded in the morning and evening) of average pain, defined as the patient-reported average pain intensity over the prior 12 hours. Percent improvement is calculated as 100 × (the weekly average of the daily average NRS pain score at week 4 - weekly average of the daily average NRS pain scores at baseline /weekly average of the daily average NRS pain scores at baseline. Patients missing a week 4 average are considered non-responders (<50% improvement or <30% improvement). The Mixed Model Repeated Measures (MMRM) model with change from baseline in the weekly average of the daily average NRS scores at week 4 as the dependent variable; week, pooled study center, treatment, and treatment by visit interaction as fixed factors, baseline weekly average of the daily average NRS scores as covariate; and patient as a random effect.
Time Frame: Baseline (day -7 to day -1), Week 4 (day 22 to day 28)
Population: Full analysis set. Participants from one site are excluded due to lack of data integrity.
Measure: Number; unit: percentage of participants
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 98 | 98 | 100
percentage of participants
  >=30% improvement from baseline | 43.9 | 43.9 | 47.0
  >=50% improvement from baseline | 22.4 | 25.5 | 28.0
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; >=30% improvement. P-value, odds ratio and CI for odds ratio are calculated using logistic model including response (yes/no) as dependent variable, treatment group and pooled study sites as factors; Test type: Superiority; p = 0.815, Regression, Logistic — 5% level of significance; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.456 to 1.856]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.893, Regression, Logistic — 5% level of significance; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.520 to 2.117]
Statistical Analysis 3: Comparison: TV-45070 4% vs Placebo; >=50% improvement. P-value, odds ratio and CI for odds ratio are calculated using logistic model including response (yes/no) as dependent variable, treatment group and pooled study sites as factors; Test type: Superiority; p = 0.430, Regression, Logistic — 5% level of significance; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.357 to 1.550]
Statistical Analysis 4: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.967, Regression, Logistic — 5% level of significance; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.494 to 2.088]

6. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in the Neuropathic Pain Symptom Inventory (NPSI) Total Score Using a Mixed Model for Repeated Measures (MMRM)
Description: NPSI is a patient-reported questionnaire to evaluate the severity of different symptoms of neuropathic pain. The questionnaire contains 10 descriptors representing 5 distinct dimensions of pain: burning pain, deep pain, paroxysmal pain, evoked pain, and paresthesia/dysesthesia, plus 2 temporal items. Descriptors are scored from 0 through 10, where higher scores represent worse pain. The total score is the sum of the scores of the 10 descriptors (Bouhassira et al 2004). The total score ranges from 0 (no pain) through 100 (worst pain imaginable). If the score for one question was missing the total score was computed as 10 times sum of scores of 9 descriptors divided by 9. If more than one question was missing then the total score was missing. Negative change from baseline scores indicated less pain.
  The MMRM used pooled study center, week, treatment, and treatment by week interaction as fixed factors and patient as a random factor.
Time Frame: Baseline (day 1 prior to dosing), Weeks 2 (day 15) and Week 4 (day 29)
Population: Full analysis set. Participants from one site are excluded due to lack of data integrity.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
units on a scale
  Baseline: number analyzed (Participants) | 98 | 98 | 100
  Baseline | 41.9 (16.45) | 44.0 (16.50) | 44.0 (15.18)
  Change from baseline at week 2: number analyzed (Participants) | 96 | 92 | 97
  Change from baseline at week 2 | -8.1 (14.13) | -9.9 (15.65) | -10.8 (14.68)
  Change from baseline at week 4: number analyzed (Participants) | 90 | 92 | 97
  Change from baseline at week 4 | -13.1 (15.76) | -14.3 (15.47) | -16.8 (17.78)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Change from baseline at Week 2 The MMRM used pooled study center, week, treatment, and treatment by week interaction as fixed factors and patient as a random factor. The unstructured covariance matrix for repeated observations within patients was used; Test type: Superiority; p = 0.251, mixed model for repeated measures — 5% level of significance; LSM of difference with placebo = 2.2, 95% CI 2-sided [-1.55 to 5.92]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; Change from baseline at Week 2. The MMRM used pooled study center, week, treatment, and treatment by week interaction as fixed factors and patient as a random factor. The unstructured covariance matrix for repeated observations within patients was used; Test type: Superiority; p = 0.495, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 1.3, 95% CI 2-sided [-2.46 to 5.07]
Statistical Analysis 3: Comparison: TV-45070 4% vs Placebo; Change from baseline at Week 4. The MMRM used pooled study center, week, treatment, and treatment by week interaction as fixed factors and patient as a random factor. The unstructured covariance matrix for repeated observations within patients was used; Test type: Superiority; p = 0.123, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 3.1, 95% CI 2-sided [-0.84 to 7.06]
Statistical Analysis 4: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p = 0.160, miex model for repeated measures — 5% level of significance; LSM difference from placebo = 2.8, 95% CI 2-sided [-1.12 to 6.77]

7. Secondary Outcome: Change From Baseline to Week 4 in the Neuropathic Pain Impact on Quality of Life (NePIQoL) Total Score
Description: NePIQoL is a questionnaire that contains 41 items to evaluate quality of life in patients with neuropathic pain. Each question has responses ranging from strongly agree or always to strongly disagree or never. Questions are scored on a 5-point scale from 1 through 5, where higher scores represent greater pain-related interference in quality of life. Total range is 41 (great quality of life) to 205 (worst quality of life). Negative change from baseline scores indicated an improving quality of life.
Time Frame: Baseline (day 1), Week 4 (day 29)
Population: Full analysis set. Participants from one site are excluded due to lack of data integrity.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
units on a scale
  Baseline: number analyzed (Participants) | 98 | 98 | 100
  Baseline | 127.1 (18.73) | 126.5 (20.36) | 127.6 (19.03)
  Change from baseline at week 4: number analyzed (Participants) | 90 | 92 | 97
  Change from baseline at week 4 | -11.5 (17.98) | 11.3 (20.09) | -12.6 (19.93)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Test type: Superiority; p = 0.609, ANCOVA — 5% level of significance; ANCOVA model includes study center, treatment, and baseline; LSM difference from placebo = 1.3, 95% CI 2-sided [-3.81 to 6.48]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; Test type: Superiority; p = 0.427, ANCOVA — 5% level of significance; ANCOVA model includes study center, treatment, and baseline; LSM difference with placebo = 2.1, 95% CI 2-sided [-3.05 to 7.19]

8. Secondary Outcome: Participants' Global Assess of Treatment as Measured by the Patient Global Impression of Change (PGIC) at Weeks 2 and 4 Using a Mixed Model for Repeated Measures (MMRM)
Description: PGIC is a standardized self-report tool that measures the change in a patient's overall status rating since the start of treatment on 7-point scale (Hurst and Bolton 2004). The 7-point scale is defined as: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse.
  The MMRM used pooled study center, week, treatment, and treatment by week interaction as fixed factors and patient as a random factor.
Time Frame: Weeks 2 (day 15) and Week 4 (day 29)
Population: Full analysis set. Participants from one site are excluded due to lack of data integrity. Data collected beyond last dose of study medication plus 3 days are excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
units on a scale
  Week 2: number analyzed (Participants) | 96 | 92 | 97
  Week 2 | 2.9 (0.87) | 2.9 (0.92) | 2.7 (0.82)
  Week 4: number analyzed (Participants) | 90 | 92 | 97
  Week 4 | 2.6 (1.08) | 2.5 (1.12) | 2.4 (1.07)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Week 2 Mixed model for repeated measures (MMRM) with pooled study center, week, treatment, and treatment by week interaction as fixed factors and patient as a random factor. The unstructured covariance matrix for repeated observations within patients was used; Test type: Superiority; p = 0.166, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.2, 95% CI 2-sided [-0.07 to 0.43]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.046, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.3, 95% CI 2-sided [0.00 to 0.51]
Statistical Analysis 3: Comparison: TV-45070 4% vs Placebo; Week 4 Mixed model for repeated measures (MMRM) with pooled study center, week, treatment, and treatment by week interaction as fixed factors and patient as a random factor. The unstructured covariance matrix for repeated observations within patients was used; Test type: Superiority; p = 0.152, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.2, 95% CI 2-sided [-0.08 to 0.53]
Statistical Analysis 4: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.342, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.1, 95% CI 2-sided [-0.16 to 0.46]

9. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in the Daily Sleep Interference Scale (DSIS) Using a Mixed Model for Repeated Measures
Description: DSIS is an 11-point scale that asks the patient to "select the number that best describes how much your pain has interfered with your sleep during the past 24 hours." Response options range from 0 (Did not interfere with sleep) to 10 (Completely interfered with sleep/unable to sleep due to pain). Negative change from baseline scores indicate improvement (lessening) of how much pain interfered with sleep.
  The MMRM used pooled study center, week, treatment, and treatment by week interaction as fixed factors and patient as a random factor.
Time Frame: Baseline (day 1 prior to dosing), Weeks 2 (day 15) and Week 4 (day 29)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
units on a scale
  Baseline: number analyzed (Participants) | 98 | 98 | 100
  Baseline | 4.5 (1.94) | 4.4 (2.26) | 4.4 (2.00)
  Change from baseline at week 2: number analyzed (Participants) | 96 | 92 | 97
  Change from baseline at week 2 | -1.1 (1.54) | -1.1 (1.99) | -1.3 (1.99)
  Change from baseline at week 4: number analyzed (Participants) | 90 | 92 | 97
  Change from baseline at week 4 | -1.4 (1.78) | -1.5 (2.16) | -1.7 (2.24)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Change from baseline at Week 2 The inferential model includes study center, week, treatment, and treatment by week interaction as the fixed factors; baseline as a covariate and unstructured variance-covariance structure in the initial model; Test type: Superiority; p = 0.311, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.2, 95% CI 2-sided [-0.22 to 0.70]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.262, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.3, 95% CI 2-sided [-0.20 to 0.73]
Statistical Analysis 3: Comparison: TV-45070 4% vs Placebo; Change from baseline at week 4 The inferential model includes study center, week, treatment, and treatment by week interaction as the fixed factors; baseline as a covariate and unstructured variance-covariance structure in the initial model; Test type: Superiority; p = 0.065, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.5, 95% CI 2-sided [-0.03 to 0.97]
Statistical Analysis 4: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.296, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.3, 95% CI 2-sided [-0.23 to 0.76]

10. Secondary Outcome: Kaplan-Meier Estimates for First Time to Reach 30% or More Sustained Improvement in Weekly Average of the Daily Average NRS Pain Scores
Description: Percent improvement is calculated as 100*(the weekly average of the daily average NRS pain score - weekly average of the daily average NRS pain scores at baseline [days -7 to -1])/weekly average of the daily average NRS pain scores at baseline. Patients who do not reach >= 30% improvement are censored at their last non-missing weekly average. Patients who reach >= 30% improvement, but the improvement is not sustained through the end of the treatment period are censored at their last non-missing weekly average. For patients who reach >= 30% improvement that is sustained through the end through the end of the of the treatment, the time >= 30% improvement is first reached is used.
Time Frame: Baseline (days -7 to -1), Week 1 (days 1-7), Week 2 (day 8-14), Week 3 (days 15-21), Week 4 (days 22-29)
Population: Full analysis set. Participants from one site are excluded due to lack of data integrity.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 98 | 98 | 100
days | NA [NA to NA] — The median and 95% CI is not estimable if the proportion of participants' with 30% improvement is less than 0.5 | NA [NA to NA] — The median and 95% CI is not estimable if the proportion of participants' with 30% improvement is less than 0.5 | NA [15.000 to NA] — The median and 95% CI is not estimable if the proportion of participants' with 30% improvement is less than 0.5
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Test type: Superiority; p = 0.245, Regression, Cox — 5% level of significance
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; Test type: Superiority; p = 0.304, Regression, Cox — 5% level of significance

11. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Maximal Intensity of Brush-Evoked Allodynia as Measured on an 11-point Numeric Rating Scale (NRS) Using a Mixed Model for Repeated Measures (MMRM)
Description: Allodynia refers to central pain sensitization (increased response of neurons) following normally non-painful, often repetitive, stimulation. In this case, pain evoked by innocuous brush is measured on an 11-point NRS where 0=no pain and 11=worst pain imaginable as reported by patients Negative change from baseline scores indicate improvement (lessening) of pain.
Time Frame: Baseline (day 1 prior to dosing), Weeks 2 (day 15) and Week 4 (day 29)
Population: Full analysis set. Participants from one site are excluded due to lack of data integrity. Participants from two other sites are excluded dince the two sites incorrectly assessed allodynia. If brush-evoked allodynia was not present at screening, it was not rechecked on subsequent visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
units on a scale
  Baseline: number analyzed (Participants) | 79 | 79 | 85
  Baseline | 1.6 (1.54) | 1.8 (2.28) | 2.0 (2.24)
  Change from baseline at week 2: number analyzed (Participants) | 54 | 47 | 62
  Change from baseline at week 2 | -0.7 (1.47) | -1.0 (2.25) | -0.8 (1.53)
  Change from baseline at week 4: number analyzed (Participants) | 53 | 46 | 62
  Change from baseline at week 4 | -0.7 (1.45) | -0.7 (2.30) | -0.7 (1.76)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.556, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = -0.1, 95% CI 2-sided [-0.61 to 0.33]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.482, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = -0.2, 95% CI 2-sided [-0.65 to 0.31]
Statistical Analysis 3: Comparison: TV-45070 4% vs Placebo; Change from baseline at week 4. The inferential model includes study center, week, treatment, and treatment by week interaction as the fixed factors; baseline as a covariate and unstructured variance-covariance structure in the initial model; Test type: Superiority; p = 0.333, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = -0.3, 95% CI 2-sided [-0.81 to 0.28]
Statistical Analysis 4: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.833, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = -0.1, 95% CI 2-sided [-0.62 to 0.50]

12. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Maximal Intensity of Punctate-Evoked Hyperalgesia as Measured on an 11-point Numeric Rating Scale (NRS) Using a Mixed Model for Repeated Measures (MMRM)
Description: Hyperalgesia refers to increased pain from a stimulus that normally provokes pain. In this case, pain is evoked by punctate skin stimulation using a Medipin® and is measured on an 11-point NRS where 0=no pain and 11=worst pain imaginable as reported by patients. Negative change from baseline scores indicate improvement (lessening) of pain.
  The MMRM used pooled study center, week, treatment, and treatment by week interaction as fixed factors and patient as a random factor. The unstructured covariance matrix for repeated observations within patients was used.
Time Frame: Baseline (day 1 prior to dosing), Weeks 2 (day 15) and Week 4 (day 29)
Population: Full analysis set. Participants from one site are excluded due to lack of data integrity. Participants from two other sites are excluded since the two sites incorrectly assessed allodynia. If punctate-evoked hyperalgesia was not present at screening, it was not rechecked on subsequent visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
units on a scale
  Baseline: number analyzed (Participants) | 79 | 79 | 85
  Baseline | 2.4 (2.03) | 3.0 (2.48) | 2.8 (2.57)
  Change from baseline at week 2: number analyzed (Participants) | 60 | 59 | 64
  Change from baseline at week 2 | -1.0 (2.02) | -1.3 (2.16) | -1.1 (1.91)
  Change from baseline at week 4: number analyzed (Participants) | 59 | 57 | 64
  Change from baseline at week 4 | -1.0 (2.08) | -1.5 (2.36) | -1.4 (2.00)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.563, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = -0.2, 95% CI 2-sided [-0.75 to 0.41]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; Change from baseline at week 2. The inferential model includes study center, week, treatment, and treatment by week interaction as the fixed factors; baseline as a covariate and unstructured variance-covariance structure in the initial model; Test type: Superiority; p = 0.804, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = -0.1, 95% CI 2-sided [-0.64 to 0.50]
Statistical Analysis 3: Comparison: TV-45070 4% vs Placebo; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.714, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.1, 95% CI 2-sided [-0.49 to 0.71]
Statistical Analysis 4: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.871, mixed model for repeated measures — 5% level of siignificance; LSM difference from placebo = 0.0, 95% CI 2-sided [-0.64 to 0.55]

13. Secondary Outcome: Participants With Treatment-Emergent Adverse Events
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: day 1 up to day 57
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 100 | 98 | 100
Participants
  Any treatment-emergent adverse event | 15 | 32 | 24
  Severe TEAE | 0 | 1 | 0
  Treatment-related TEAE | 5 | 10 | 11
  Deaths | 0 | 0 | 0
  Serious TEAE | 0 | 1 | 0
  Withdrawn from treatment due to TEAE | 4 | 4 | 3

ADVERSE EVENTS:
Time Frame: day 1 up to day 57
Groups:
- TV-45070 (8%): TV-45070 ointment in a 8% strength applied topically twice daily to the area of postherpetic neuralgia (PHN) pain during the treatment period from days 1 through 28.
Arm/Group | TV-45070 4% | TV-45070 (8%) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/98 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/98 | 0/100
Other Adverse Events (participants affected / at risk) | 2/100 | 5/98 | 1/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TV-45070 4% (N=100) | TV-45070 (8%) (N=98) | Placebo (N=100)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TV-45070 4% (N=100) | TV-45070 (8%) (N=98) | Placebo (N=100)
Application site erythema (General disorders) | 2 (3) | 5 (5) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02365636/Prot_001.pdf
  • Statistical Analysis Plan (2015-09-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT02365636/SAP_000.pdf